CLINICAL TRIAL: NCT02216253
Title: L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract to Prevent Postoperative Urinary Tract Infection: a Double-blind Randomized Controlled Trial.
Brief Title: L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract to Prevent Postoperative Urinary Tract Infection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Umberto Leone Roberti Maggiore, MD, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UTI 2014
Record Dates: First submitted 2014-08-09; First posted 2014-08-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Urinary Tract Infection; Pelvic Organ Prolapse; Urinary Incontinence
Keywords: Urinary tract infection; Pelvic organ prolapse; Urinary incontinence; Stress urinary incontinence; Mixed Urinary incontinence; L-methionine; Placebo
MeSH Terms: conditions — Urinary Tract Infections; Pelvic Organ Prolapse; Urinary Incontinence; Urinary Incontinence, Stress | interventions — Methionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract (Active Comparator): The combination of L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract will be administered in tablet twice a day 7 days before and after surgery
  Interventions: Drug: L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract
- Placebo (Placebo Comparator): Placebo tablet twice a day 7 days before and after surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract — L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract tablet twice a day 7 days before and after surgery
  Arms: L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract
Other: Placebo — Placebo tablet twice a day 7 days before and after surgery
  Arms: Placebo

SUMMARY:
This study will include women who will undergo pelvic reconstructive surgery and/or anti-incontinence sling procedures. Patients will be randomized to the combination of L-methionine, Hibiscus Sabdariffa and Boswellia Leaf Extract in tablet or placebo twice a day during the seven days before and after surgery (total of 14 days). In this randomized, double-blind study, the investigators will assess treatment of clinically suspected or culture-proven urinary tract infections within 3 weeks of surgery (primary outcome), and risk factors for treatment for postoperative urinary tract infections (secondary outcomes) between the two study groups.

ELIGIBILITY:
Inclusion Criteria:

* postoperative transurethral catheterization after surgery for pelvic organ prolapse and/or urinary incontinence
* patients aged ≥ 18 years

Exclusion Criteria:

* acute urinary tract infection at the moment of inclusion in the study
* antibiotic treatment prescribed for any other cause than urinary tract infection
* pregnancy
* known allergy to one of the elements of the active compound
* surgery for mesh excision
* surgery for urethral diverticulum
* surgery for fistula repair
* surgery for sacral neuromodulation
* any condition precluding the acquisition of written consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Treatment for urinary tract infection after surgery. | 3 weeks after surgery.
  To assess any treatment received for clinically suspected or culture-proven urinary tract infection within 3 weeks of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Leone Roberti Maggiore, MD, Principal Investigator — IRCCS San Raffaele Hospital and Vita-Salute San Raffaele University; Stefano Salvatore, MD, Study Director — IRCCS San Raffaele Hospital and Vita-Salute San Raffaele University
Locations (1):
- IRCCS San Raffaele Hospital and Vita-Salute San Raffaele University, Milan, Lombardy, Italy